CLINICAL TRIAL: NCT00358488
Title: A Multi-enter, Randomized, Double-blind, Placebo-controlled, Four-way Incomplete Block Crossover Study to Examine Efficacy, Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single and Repeat Administration of Three Inhaled Doses (10, 15, and 20 mcg) of GSK159797
Brief Title: Study Investigating Repeat Doses Of A New Medication (GSK159797) In Asthmatic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2E106359
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Safety; Asthmatic patients; GSK159797; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- GSK159797 (10, 15, and 20mcg) (Experimental): GSK159797 (10, 15, and 20mcg)
  Interventions: Drug: GSK159797 (10, 15, and 20mcg)
- salbutamol (Experimental): salbutamol
  Interventions: Drug: salbutamol
- salmeterol 50mcg (Experimental): salmeterol 50mcg
  Interventions: Drug: salmeterol 50mcg
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GSK159797 (10, 15, and 20mcg) — GSK159797 (10, 15, and 20mcg)
  Arms: GSK159797 (10, 15, and 20mcg)
Drug: salbutamol — salbutamol
  Arms: salbutamol
Drug: salmeterol 50mcg — salmeterol 50mcg
  Arms: salmeterol 50mcg
Drug: placebo — placebo
  Other Names: GSK159797 (10; 15; and 20mcg); salbutamol; salmeterol 50mcg
  Arms: placebo

SUMMARY:
This study is designed to determine the efficacy and safety of a new long-acting beta-agonist for asthma patients (GSK159797) following dosing for 14 days.

ELIGIBILITY:
Inclusion criteria:

* Subjects with documented history of persistent asthma using corticosteroids at a total daily dose of 200 to 200mcg of FP or equivalent corticosteroid
* Female subjects only using acceptable birth control method
* Non-smokers
* FEV1 between 60 and 90% predicted
* Increase in FEV1 12% or greater and 300mL and greater after salbutamol use

Exclusion criteria:

* Past or present disease conditions
* Normal screening Holter ECG
* Respiratory tract infection within 4 weeks of screening
* History of life threatening asthma
* Previous use of COA

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in trough FEV1 | after 14 day repeat doses

SECONDARY OUTCOMES:
Mean change from baseline in trough FEV1 | after a single dose
Mean change from baseline in trough FEV1 | after 7 days repeat dosing
Change from baseline in weighted mean FEV1 0-2 hours, 0-4 hours, 0-24 hours | Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- Germany (2):
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Berlin, State of Berlin
- GSK Investigational Site, Utrecht, Netherlands
- GSK Investigational Site, Moscow, Russia
- GSK Investigational Site, Lund, Sweden
- GSK Investigational Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2E106359 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register